CLINICAL TRIAL: NCT00240318
Title: A 104-Week, Open-label, Multi-centre, Phase IIIb Study Evaluating the Effect of Treatment With Rosuvastatin 40 mg on Atherosclerotic Disease as Measured by Intravascular Ultrasound and Quantitative Coronary Angiography in Subjects Undergoing Coronary Angiography Who Have Coronary Artery Disease
Brief Title: A Study To Evaluate the Effect of Rosuvastatin On Intravascular Ultrasound-Derived Coronary Atheroma Burden (ASTEROID)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3562C00076
Record Dates: First submitted 2005-10-16; First posted 2005-10-18 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Coronary Arteriosclerosis
Keywords: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: Rosuvastatin calcium
  Other Names: Crestor

SUMMARY:
The purpose of this study is to see if 40 mg of rosuvastatin taken daily will reduce the atherosclerosis (fatty deposits) in your arteries

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for coronary catheterization. Target Coronary Artery: The target vessel must have .50% reduction in lumen diameter by angiographic visual estimation throughout a segment of at least 40 mm in length (the target segment) and the vessel must be large enough to accommodate the IVUS catheter. A lesion of up to 60% is permitted distal to the target segment. Side branches of the target (imaged) vessel may be narrowed up to 70% by visual estimation, provided the target segment contains no lesion greater than 50%.

Exclusion Criteria:

Use of lipid-lowering medication for more than 3 months within the previous 12 months. Longer periods of treatment are not permitted because of the potential effects of such therapy on coronary atherosclerosis. Subjects receiving treatment with a lipid-lowering medication within the past 4 weeks require a 4-week wash-out period following which a baseline lipid profile will be taken at visit 2.

Clinically significant heart disease which, in the opinion of the Principal Investigator (or designee), is likely to require coronary bypass surgery, cardiac transplantation, surgical repair and/or replacement during the course of the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2002-11; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
to evaluate whether 2 years of treatment with 40 mg rosuvastatin results in regression of coronary artery atheroma burden via the total atheroma volume in the most diseased segment or the percent atheroma volume, as measured by IVUS

SECONDARY OUTCOMES:
to evaluate whether treatment with rosuvastatin results in:
Regression of coronary artery atheroma burden, as assessed by TAV
Regression of coronary artery disease as measured by quantitative coronary angiography (QCA).
To evaluate the change in lipid and lipoprotein levels as assessed by percentage change from baseline.
To evaluate the safety of rosuvastatin

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Crestor Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (61):
- United States (24):
  - Research Site, Birmingham, Alabama
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Santa Rosa, California
  - Research Site, Stockton, California
  - Research Site, Denver, Colorado
  - Research Site, Hartford, Connecticut
  - Research Site, Atlantis, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Auburn, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Petoskey, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Buffalo, New York
  - Research Site, Valhalla, New York
  - Research Site, Williamsville, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Toledo, Ohio
  - Research Site, Danville, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, Milwaukee, Wisconsin
- Australia (4):
  - Research Site, Auchenflower
  - Research Site, Clayton
  - Research Site, Heidelberg
  - Research Site, New Lambton
- Belgium (4):
  - Research Site, Aalst
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Liège
- Canada (3):
  - Research Site, Halifax, Nova Scotia
  - Research Site, Montreal, Quebec
  - Research Site, Ste-Foy, Quebec
- France (8):
  - Research Site, Créteil
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Massy
  - Research Site, Melun
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Toulouse
- Italy (9):
  - Research Site, Rozzano, Milan
  - Research Site, Mirano, Venezia
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Pavia
  - Research Site, Pisa
  - Research Site, Rome
  - Research Site, Siena
  - Research Site, Udine
- Netherlands (4):
  - Research Site, Amsterdam
  - Research Site, Maastricht
  - Research Site, Nieuwegein
  - Research Site, Zwolle
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Murias
  - Research Site, Valladolid

REFERENCES:
- [Result] Nissen SE, Nicholls SJ, Sipahi I, Libby P, Raichlen JS, Ballantyne CM, Davignon J, Erbel R, Fruchart JC, Tardif JC, Schoenhagen P, Crowe T, Cain V, Wolski K, Goormastic M, Tuzcu EM; ASTEROID Investigators. Effect of very high-intensity statin therapy on regression of coronary atherosclerosis: the ASTEROID trial. JAMA. 2006 Apr 5;295(13):1556-65. doi: 10.1001/jama.295.13.jpc60002. Epub 2006 Mar 13. PMID 16533939